CLINICAL TRIAL: NCT00768001
Title: Genetic Analysis of Liver Cancer
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: Samuel So (Other)
Responsible Party: Sponsor-Investigator, Samuel So, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Other Study IDs: HEP0012; 98717 (Other: SU)
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Liver Cancer; Hepatitis B; Hepatitis C; Hepatobiliary Cancers; Hepatobiliary Cancers Liver
MeSH Terms: conditions — Liver Neoplasms; Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor sample

SUMMARY:
Liver cancer is a leading cause of cancer deaths worldwide. While the molecular pathogenesis of liver cancer has been extensively studied, less is known about how the molecular biology of liver cancer influences clinical outcome and treatment response. We are developing a translational research program that will characterize molecular changes in liver cancer. We plan to use molecular information obtained from studying liver tumor tissues to develop new diagnostics and treatment regimens for patients with these cancers. The experimental approach will require freezing fresh tumor tissues obtained from surgical procedures, which will be subsequently used for analysis of DNA, protein and mRNA expression. Many patients with liver cancer are referred to the Stanford Liver Tumor Board for consultation and treatment recommendations. We propose to gather tissue samples from those who subsequently undergo biopsy, liver resection surgery, or transplant surgery.

ELIGIBILITY:
Inclusion Criteria:3.1.1 Male or female patients 18 years of age and above. 3.1.2 Patients diagnosed with liver cancer based on biopsy or serum alpha-fetoprotein level, associated with characteristic hypervascular liver tumors on triphasic spiral CT scan or MRI. Patients with non-cancer liver conditions such as cirrhosis, adenoma, cholangioma, or nodular hyperplasia. Patients with metastatic tumor from anther organ, such as metastatic colon cancer.

3.13 Ability to understand and the willingness to sign a written informed consent document. Exclusion Criteria:3.2.1Female patients who are pregnant or nursing will be excluded from the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel So, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States